CLINICAL TRIAL: NCT02667769
Title: Comparison of Two Protocols on the Implementation of a Fasting Day to Check the Basal Insulin Replacement in Type 1 Diabetes: Complete Fasting Compared to the Permission for Carbohydrate- and Calorie-free Food
Brief Title: Comparison of Two Protocols on the Implementation of a Fasting Day in Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diabeteszentrum Bad Lauterberg im Harz (Other)
Responsible Party: Principal Investigator, Michael A. Nauck, Prof. Dr. med. Michael A. Nauck, Diabeteszentrum Bad Lauterberg im Harz
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DZBL-2014-2
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting day without any food (Other): Complete fasting: On a fast day under this Protocol no solid food may be eaten unless it is solid, medically prescribed part of a bedtime snack just before falling asleep (which must sometimes be to prevent nocturnal hypoglycaemia with injection of basal insulin before going to sleep) , Otherwise, the patient have ad libitum access to mineral water and unsweetened tea (possibly a fluid intake restriction should be considered for other diseases).
  Interventions: Other: Fasting day
- Fasting day with calorie- & carbohydrate-free food (Other): During a fasting day for this protocol, patients may calories in unlimited quantity and (with calorie-free dressing) Take carb food like tomatoes, cucumbers, lettuce to be, both during meal periods and in between, if desired.
  Interventions: Other: Fasting day

INTERVENTIONS:
Other: Fasting day — A day of fasting started at 18.00 clock with a blood glucose test and is only started when on the same day no significant hypoglycemia (blood glucose <55 mg / dl) occurred, and when at 18.00 clock the blood sugar in the defined target range (70-180 mg / dl) is. Carried out during the fasting day standardized blood samples for measurement of plasma glucose with an appropriate laboratory method at 18.00, 20:00, 22:00, 12:00, 2:00, 4:00, 6:45, 9:00, 12:00, 14:00 and again at 18.00 clock. Because the determination of plasma glucose in the laboratory will take some time, is always for guidance and also measured with a fast measurement method, in order to treat at high levels of blood sugar with additional insulin correction, and to treat hypoglycaemia low blood sugar or to prevent hypoglycaemia.

SUMMARY:
This is a prospective study with a "crossover design", where fasting with a day of complete fasting and a fasting day with the permission intake of calories- and carbohydrate-free foods are compared in a randomized order. Underlying hypothesis is that at the same basal insulin substitution with the fasting of both protocols , no significant differences in the glucose-day or -night profiles revealed. So the same conclusions regarding the "consistency" of basal insulin dosing revealed during the implementation of the part of patients is rated as more pleasant when calories and carbohydrates-free food are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Basal insulin substitution with neutrales Protamin Hagedorn (NPH) -insulin (at least twice a day), insulin detemir (twice a day), insulin glargine (once or twice a day) or with insulin pump
* Diabetes duration > 2 years
* Body-mass-index between 19 and 35 kg/m², including
* written consent

Exclusion Criteria:

* No pregnancy in woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma glucose day- and night profiles | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haase M, Kahle M, Janert M, Meier JJ, Nauck MA. Basal rate tests (24-hour fasts) performed in type-1 diabetic subjects with either absolute fasting or snacks containing negligible carbohydrate amounts result in similar glucose profiles: A randomized controlled prospective trial. Diabetes Obes Metab. 2017 Jun;19(6):783-790. doi: 10.1111/dom.12868. Epub 2017 Mar 20. PMID 28058800